CLINICAL TRIAL: NCT04904185
Title: Adoptive Transfer of ImmPACT Expanded Multiple Antigen Specific Endogenously Derived T Cells (MASE-T) in Combination With Lymphodepletion and Anti-PD-1 to Patients With Metastatic Melanoma
Brief Title: ImmPACT Expanded Multiple Antigen Specific Endogenously Derived T Cells (MASE-T) to Patients With Metastatic Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Evaluation of step A did not support addition of pembrolizumab in step B
Sponsor: Inge Marie Svane (Other)
Collaborators: Technical University of Denmark (Other)
Responsible Party: Sponsor-Investigator, Inge Marie Svane, M.D., Professor, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MM2011
Record Dates: First submitted 2021-05-22; First posted 2021-05-27 (Actual); Results first posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Malignant Melanoma
Keywords: Adoptive Cell Therapy; Immune Therapy; Multiple Antigen Specific Endogenously derived T cells
MeSH Terms: conditions — Melanoma | interventions — Cyclophosphamide; fludarabine phosphate; pembrolizumab

STUDY DESIGN:
Intervention Model Description: 12 Patients will be indluced in two steps.
  * Part A (6 patients): Lymphodepleting chemotherapy (cyclophosphamide 500 mg/m2/day i.v. on day -4, -3, -2 and fludarabine 30 mg/m2/day i.v. on day -4, -3) followed by i.v. infusion of the MASE-T product on day 0. If the production of the MASE-T cell product was feasible for the majority (>50%) of patients intended to treat in Arm A and the toxicity was acceptable, six patients will further be included in part B.
  * Part B (6 patients): Lymphodepleting chemotherapy (cyclophosphamide 500 mg/m2/day i.v. on day -4, -3, -2 and fludarabine 30 mg/m2/day i.v on day -4, -3) followed by i.v infusion of the MASE-T product on day 0. Pembrolizumab 2 mg/kg will be administered on day -1 and day +21.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A (Other): Six patients will be included in Part A. After inclusion 300 mL blood will be drawn from the patients for the production of the MASE-T cell product. Four days prior to MASE-T infusion the patient will receive lymphodepleting chemotherapy (cyclophosphamide 500 mg/m2/day i.v. on day -4, -3, -2 and fludarabine 30 mg/m2/day i.v. on day -4, -3) followed by i.v. infusion of the MASE-T product on day 0.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Biological: Multiple Antigen Specific Endogenously derived T cells
- Part B (Other): Six patients will be includede in Part B. After inclusion 300 mL blood will be drawn from the patients for the production of the MASE-T cell product. Four days prior to MASE-T infusion the patient will receive lymphodepleting chemotherapy (cyclophosphamide 500 mg/m2/day i.v. on day -4, -3, -2 and fludarabine 30 mg/m2/day i.v on day -4, -3) followed by i.v infusion of the MASE-T product on day 0. Pembrolizumab 2 mg/kg will be administered on day -1 and day +21.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Biological: Multiple Antigen Specific Endogenously derived T cells; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide 500 mg/m2 is administered i.v. on day -4, -3 and -2
Drug: Fludarabine Phosphate — Fludarabine Phosphate 30 mg/m2 is administered on day -4 and -3
Biological: Multiple Antigen Specific Endogenously derived T cells — Antigen specific, ex vivo expanded T cells derived from peripheral blood T cells
  Other Names: MASE-T
Drug: Pembrolizumab — Pembrolizumab 2 mg/kg is administered on day -1 and on day 21. The medicine is administered over 30 minutes
  Arms: Part B

SUMMARY:
With the introduction of checkpoint inhibitors substantial improvements have been made in the treatment of malignant melanoma (MM). Despite this still a a subset of patients, approximately 50 %, experience no response to therapy.

One of the strategies to overcome these obstacles have been ACT with tumour infiltrating lymphocytes (TILs). Most TIL based ACT products are non-specifically expanded providing growth preference to co-infiltrated virus specific T cells, and it is currently challenging to expand T cells in an antigen-specific manner, while at the same time obtaining the ideal functional characteristics for specific and strong tumour-killing capacity with sufficient persistence.

In this phase I trial artificial antigen-presenting scaffolds for antigen-driven T cell expansion are used. These scaffolds will generate a MASE-T cell product enriched for selected specificities towards antigens known to be expressed by melanoma cells The aim of the study is to demonstrate that treatment with af MASE-T cell product i safe and feasible. Further the study will elucidate whether treament with the MASE-T cell product leads to objective responses and improves progression free survival (PFS).

DETAILED DESCRIPTION:
There are around 350-400 new cases of patients with metastatic melanoma (MM) per year in Denmark. MM is a very aggressive cancer with a poor prognosis. Traditional oncological treatments such as surgery, chemotherapy and radiation therapy have a poor effect, and the 5-year overall survival has hitherto been less than 10 %.Substantial improvements have been made in the treatment of MM; especially immunotherapy is showing promising results with checkpoint inhibitors (CPI) such as programmed cell death protein 1 (PD-1) and Cytotoxic T Lymphocyte-associated Antigen 4 (CTLA-4) blocking antibodies administered as standard treatment in the frontline. The 5-year overall survival has now reached 52 %, 44 % and 26 % in nivolumab/ipilimumab, nivolumab, and ipilimumab respectively. However, a subset of patients - approximately 50 % experience no response to therapy, with clear primary resistance. One of the strategies to overcome these obstacles have been ACT with tumour infiltrating lymphocytes (TILs). A crucial condition for optimal ACT based on TILs is the generation of sufficient numbers of tumourreactive T cells. However, the expansion of TILs requires extensive ex vivo culturing often at the cost of T cell differentiation and functional activity. Most TIL based ACT products are non-specifically expanded providing growth preference to co-infiltrated virus specific T cells, and it is currently challenging to expand T cells in an antigen-specific manner, while at the same time obtaining the ideal functional characteristics for specific and strong tumour-killing capacity with sufficient persistence. Recent data suggest that the majority of tumour specific T cells responsible for tumour rejection under CPI are recruited from peripheral blood and lymph system, while not present in the tumour prior to treatment. This is supported by the finding that most tumour resident T cells are dysfunctional.

To overcome the current limitations in the treatment of malignant melanoma artificial antigen-presenting scaffolds for antigen-driven T cell expansion, generating a MASE-T cell product enriched for selected specificities towards antigens known to be expressed by melanoma cells has been designed. The antigen-scaffolds will ensuring optimal T cell stimulation by mimicking the in vivo stimulation of T cells by dendritic cells in the lymph nodes. The scaffolds contain both the antigen specific element - in the form of a peptide-MHC molecule and cytokine (IL2 and IL21), to provide growth and functional signals to the antigen specific T cell. As a result of this T cell expansion strategy, we can obtain a T cell product enriched for tumourantigen specific T cells. Superior functional activity towards tumor cells and antigen recognition compared to conventional T cell expansion strategies has been demonstrated in-vitro. Importantly, antigen-specific T cells in the MASE-T cell product possess a 'younger' phenotype, which has previously been described to correlate with improved in vivo persistence.

The study is a phase 1, non-randomized study. The trial will be conducted in two parts (A and B). Patients will be treated as followed:

* Part A (6 patients): Lymphodepleting chemotherapy (cyclophosphamide 500 mg/m2/day i.v. on day -4, -3, -2 and fludarabine 30 mg/m2/day i.v. on day -4, -3) followed by i.v. infusion of the MASE-T product on day 0. If the production of the MASE-T cell product was feasible for the majority (≥50%) of patients intended to treat in Arm A and the toxicity was acceptable, six patients will further be included in part B.
* Part B (6 patients): Lymphodepleting chemotherapy (cyclophosphamide 500 mg/m2/day i.v. on day -4, -3, -2 and fludarabine 30 mg/m2/day i.v on day -4, -3) followed by i.v infusion of the MASE-T product on day 0. Pembrolizumab 2 mg/kg will be administered on day -1 and day +21.

The primary objective is to evaluate the safety and feasibility of the MASE-T treatment alone or in combination with Pembrolizumab in patients with stage IV metastatic melanoma according to Common Terminology Criteria for Adverse Events (CTCAE version 5.0).

The secondary objectives are to evaluate T cell profile and persistence in vivo from tumor biopsies and blood samples as well as evaluation of the clinical efficacy of the treatment according to RECIST 1.1 and iRECIST. In addition, best overall response (BOR), duration of response (DOR), overall survival (OS), progression-free survival (PFS) will be monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 ≤ 75
2. Progressive disease on or after anti-PD-1/anti-PD-L1 monotherapy or progressive disease on or after anti PD-1 plus anti-CTLA-4 therapy
3. The patient has histologically confirmed metastatic melanoma
4. HLA-A2 positive
5. At least one measurable parameter according to RECIST version 1.1 guidelines
6. ECOG performance status of 0 or 1
7. No significant toxicity from previous cancer treatments (CTC ≤ 1)
8. Women of childbearing potential: Negative serum pregnancy test and must use effective contraception. This applies from screening and until 6 months after treatment. Birth control pills, spiral, depot injection with gestagen, subdermal implantation, hormonal vaginal ring and transdermal depot patch are all considered effective contraceptives
9. Men with female partner of childbearing potential must use effective contraception from screening and until 6 months after treatment. Effective contraceptives are as described above for the female partner. In addition, documented vasectomy and sterility or double barrier contraception are considered effective contraceptives
10. Signed statement of consent after receiving oral and written study information
11. Willingness to participate in the planned treatment and follow-up and capable of handling
12. The patient has met the following haematological and biochemical criteria:

    1. AST and ALT ≤2,5 X ULN or ≤5 X ULN with liver metastases
    2. Serum total bilirubin ≤1,5 X ULN or direct bilirubin ≤ ULN for patient with total bilirubin level > 1,5 ULN
    3. Serum creatinine ≤1,5 X ULN
    4. ANC (Absolute Neutrophil Count) ≥1,000/mcL
    5. Platelets ≥ 75,000 /mcL
    6. Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L

Exclusion Criteria:

1. Another malignancy or concurrent malignancy unless disease-free for 3 years
2. Requirement for immunosuppressive doses of systemic corticosteroids (>10 mg/day prednisone or equivalent) or other immunosuppressive drugs within the last 3 weeks prior to screening
3. Prior treatment with adoptive transfer of Tumor Infiltrating T cells (TIL)
4. Grade 3-4 adverse events upon treatment with PD-1 checkpoint inhibitors (only phase B)
5. The patient has CNS metastases and/or carcinomatous meningitis
6. The patient has any condition that will interfere with patient compliance or safety (including but not limited to psychiatric or substance abuse disorders)
7. The patient is pregnant or breastfeeding
8. The patient has an active infection requiring systemic therapy
9. The patient has received a live virus vaccine within 30 days of planned start of therapy
10. Significant medical disorder according to investigator; e.g severe asthma or chronic obstructive lung disease, dysregulated heart disease or dysregulated diabetes mellitus.
11. Concurrent treatment with other experimental drugs
12. Any significant active autoimmune disease
13. Severe allergy or anaphylactic reactions earlier in life
14. Known hypersensitivity to one of the active drugs or one or more of the excipients.
15. Unrelieved lower urinary tract obstruction

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Inge M Svane, Prof., M.D., Study Director — Study Director, National Center for Cancer Immune Therapy, Depth of Oncology, Herlev Hospital; Tine J Monberg, M.D., Principal Investigator — Ph.d. student, National Center for Cancer Immune Therapy, Depth of Oncology, Herlev Hospital
Locations (1):
- National Center for Cancer Immune Therapy (CCIT-DK), Herlev, Denmark

RESULTS

PARTICIPANT FLOW:
Groups:
- Part B: No patients enrolled due to premature closure of the trial
Period: Overall Study
Arm/Group | Part A | Part B
Started | 8 | 0
Completed | 6 | 0
Not Completed | 2 | 0
Not completed — Expansion failure | 1 | 0
Not completed — Late response on prior treatment | 1 | 0

BASELINE CHARACTERISTICS:
Population: No patients were enrolled in part B due to premature closure of the trial
Groups:
- Part A: Six patients were included in Part A. After inclusion 300 mL blood will be drawn from the patients for the production of the MASE-T cell product. Four days prior to MASE-T infusion the patient will receive lymphodepleting chemotherapy (cyclophosphamide 500 mg/m2/day i.v. on day -4, -3, -2 and fludarabine 30 mg/m2/day i.v. on day -4, -3) followed by i.v. infusion of the MASE-T product on day 0.
  Cyclophosphamide: Cyclophosphamide 500 mg/m2 is administered i.v. on day -4, -3 and -2
  Fludarabine Phosphate: Fludarabine Phosphate 30 mg/m2 is administered on day -4 and -3
  Multiple Antigen Specific Endogenously derived T cells: Antigen specific, ex vivo expanded T cells derived from peripheral blood T cells
- Total: Total of all reporting groups
Arm/Group | Part A | Part B | Total
Number analyzed (Participants) | 6 | 0 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 0 | 4
  >=65 years | 2 | 0 | 2
Age, Continuous [Median (Full Range); unit: years] | 61 [28 to 75] |  | 61 [28 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 2 | 0 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
HLA-A2*02:01 positive assessed by flow cytometry [Number; unit: participants] — HLA-A2*02:01 was assessed using flow cytometry which was performed on a single blood test. Positive results were later confirmed by polymerase chain reaction (PCR)
  participants | 6 |  | 6
TET+ T cells in peripheral blood assessed by flow cytometry [Number; unit: participants] | 6 |  | 6
Performance status according to ECOG Performance Status Scale [Number; unit: participants] — ECOG Performance status:
  0: Fully active; no performance restrictions.
  1. Strenuous physical activity restricted; fully ambulatory and able to carry out light work.
  2. Capable of all self-care but unable to carry out any work activities. Up and about >50% of waking hours.
  3. Capable of only limited self-care; confined to bed or chair >50% of waking hours.
  4. Completely disabled; cannot carry out any self-care; totally confined to bed or chair.
  participants
    ECOG PS 0 | 5 |  | 5
    ECOG PS 1 | 1 |  | 1
Number of prior treatment lines [Median (Full Range); unit: lines of prior treatment] | 3.5 [1 to 4] |  | 3.5 [1 to 4]

OUTCOME MEASURES:

1. Primary Outcome: Tolerability of the Treatment
Description: Number of patients experiencing grade III or worse adverse events. The grading of adverse events was performed according to CTCAE ver. 5.0.
Time Frame: Through study completion, up to 2.8 years from begin of study
Population: No patients were enrolled in part B due to premature closure of the trial
Measure: Count of Participants; unit: Participants
Groups:
- Part A: Multiple Antigen Specific endogenously derived T cells: After inclusion 300 mL blood will be drawn from the patients for the production of the MASE-T cell product ex vivo. Four days prior to MASE-T infusion the patient will receive lymphodepleting chemotherapy (cyclophosphamide 500 mg/m2/day i.v. on day -4, -3, -2 and fludarabine 30 mg/m2/day i.v. on day -4, -3) followed by i.v. infusion of the MASE-T product on day 0.
  Cyclophosphamide: Cyclophosphamide 500 mg/m2 is administered i.v. on day -4, -3 and -2
  Fludarabine Phosphate: Fludarabine Phosphate 30 mg/m2 is administered on day -4 and -3
  Multiple Antigen Specific Endogenously derived T cells: Antigen specific, ex vivo expanded T cells derived from peripheral blood T cells
Arm/Group | Part A | Part B
Number analyzed (Participants) | 6 | 0
Participants | 6 | 0

2. Primary Outcome: Number of Patients Excluded Due to Feasibility Issues
Description: Number of patients excluded due to treatment related feasibility issues compared to the number of patients enrolled in the study.
Time Frame: Through study completion, up to 2.8 years from begin of study
Population: No patients were enrolled in part B due to premature closure of the trial
Measure: Count of Participants; unit: Participants
Groups:
- Part B: Six patients were plan for part B with the addition of of the PD-1 inhibitor Pembrolizumab. Due to delivery problems with the scaffolds the trial was, however, terminated prematurely (after Part A)
Arm/Group | Part A | Part B
Number analyzed (Participants) | 8 | 0
Participants | 1 |

3. Primary Outcome: Number of Patients Excluded Due to Safety Issues
Description: Number of patients excluded due to treatment related safety issues compared to the number of patients enrolled in the study.
Time Frame: Through study completion, up to 2.8 years from begin of study
Population: No patients were enrolled in part B due to premature closure of the trial
Measure: Count of Participants; unit: Participants
Groups:
- Part B: No patients were enrolled in part B due to premature closure of the trial
Arm/Group | Part A | Part B
Number analyzed (Participants) | 8 | 0
Participants | 0 |

4. Secondary Outcome: Best Overall Response (BOR)
Description: Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1) assessed by CT scan.
  Complete Response (CR): Disappearance of all target lesions Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions Progressive disease: >= 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions Stable disease: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study
Time Frame: The patients were evaluated every 6-12 weeks until study completion (minimum: 43 days, median: 69 days, maximum: 128 days)
Population: No patients included in part B due to premature closure of the trial
Measure: Count of Participants; unit: Participants
Arm/Group | Part A | Part B
Number analyzed (Participants) | 6 | 0
Participants
  Stable disease | 3 |
  Progressive disease | 3 |

ADVERSE EVENTS:
Time Frame: The data was collected throughout the duration of the clinical trial, from September 2021 (enrollment of the first patient) and until exclusion of the last patient in June 2024 (2.8 years) Adverse events were collected every 6-12 weeks until study completion. For the individual patient, the reporting started at the study enrolment and ended with study exclusion (median 69 days, maximum 128 days from MASE-T infusion).
Description: Serious adverse events also included AEs that:
  * Resulted in persistent or significant disability or incapacity;
  * Led to a congenital anomaly or birth defect;
  * Was a significant medical event.
  * Resulted in the transmission of an infectious agent
  * Pregnancy must follow the same transmission timing and process used for SAEs.
  A specific list of events that should not be reported is included in the protocol
Arm/Group | Part A | Part B
All-Cause Mortality (participants affected / at risk) | 5/6 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/0
Other Adverse Events (participants affected / at risk) | 6/6 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A (N=6) | Part B (N=0)
Dizziness and palor (General disorders) | 1 (1) | 0 (0)
Neutropenia (Immune system disorders) | 4 (4) | NA
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | NA
Anemia (Blood and lymphatic system disorders) | 6 (21) | NA
Diarrhea (Gastrointestinal disorders) | 1 (1) | NA
Dry mouth (General disorders) | 2 (3) | NA
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | NA
Fatique (General disorders) | 6 (19) | NA
Fever (General disorders) | 1 (1) | NA
Hyponatriemia (Metabolism and nutrition disorders) | 1 (1) | NA
Increase in CRP (General disorders) | 1 (1) | NA
Loss of appetite (Gastrointestinal disorders) | 1 (1) | NA
Lymphopenia (Immune system disorders) | 6 (12) | NA
Nausea (Gastrointestinal disorders) | 3 (3) | NA
Obstipation (Gastrointestinal disorders) | 1 (1) | NA
Pain (General disorders) | 2 (3) | NA
Trombocytopenia (Blood and lymphatic system disorders) | 2 (9) | NA
Vomiting (Gastrointestinal disorders) | 1 (1) | NA

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-27): https://cdn.clinicaltrials.gov/large-docs/85/NCT04904185/Prot_SAP_000.pdf